CLINICAL TRIAL: NCT04027335
Title: Use of the Leva Pelvic Digital Health System in Women With Fecal Incontinence: a Pilot Study
Brief Title: Use of the Leva Pelvic Digital Health System in Women With Fecal Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renovia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REN-17
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Women
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Leva Arm (Experimental): Subjects will undergo training in the use of a vaginal device and its associated app, to be used twice daily to perform pelvic floor muscle exercises guided by the device/app for 10 weeks.
  Interventions: Device: leva

INTERVENTIONS:
Device: leva — Vaginal device used for pelvic floor muscle exercises

SUMMARY:
Pilot study to understand the impact of a digital health system, including a phone app and a vaginal probe to treat fecal incontinence in women

DETAILED DESCRIPTION:
Subjects meeting inclusion/exclusion criteria at screening will complete training in behavioral therapy for the treatment of fecal incontinence and training in the use of the Leva pelvic digital health system.

Subjects will then participate in 10 weeks of at home pelvic floor muscle training using the leva device twice daily for 2 ½ minutes of training.

Adherence to the training protocol will be observed digitally, and subjects will receive phone calls every other week from research assistants reviewing their adherence.

Subjects are expected to participate in at least 80% of the weekly exercises (11 weekly).

Subjects will return to clinic at 5- and 10-weeks during the study to complete questionnaires. At 5-weeks, subjects will review the use of the device with the study assistant, who will answer any questions and repeat training if the subject desires additional training.

Following 10 weeks of training, subjects will be free to pursue any additional therapies, but will also retain the leva device and may continue its use if desired. Adherence will be monitored for one additional year, with follow up surveys to be completed by mail or digitally at 6- and 12-months

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Fecal incontinence defined as any uncontrolled loss of liquid or solid fecal material that occurs at least monthly over the last 3 months that is bothersome enough to desire treatment
3. Ambulatory

Exclusion Criteria:

1. Absence of a vagina
2. Stool consistency over the last 3 months that includes items 1 or 7 based on the Bristol Stool form scale (severe constipation or diarrhea)
3. Current or past diagnosis of colorectal or anal malignancy
4. Diagnosis of inflammatory bowel disease
5. Current or history of rectovaginal fistula or cloacal defect
6. Rectal prolapse (mucosal or full thickness)
7. Prior removal or diversion of any portion of colon or rectum
8. Prior pelvic floor or abdominal radiation
9. Refusal or inability to provide written consent
10. Inability to utilize smart phone technology ("app" use)
11. Fecal impaction by exam
12. Stage 3 or 4 pelvic organ prolapse
13. Incontinence only to flatus
14. Supervised anal sphincter exercise/pelvic floor muscle training with or without biofeedback currently or within the past 6 months.
15. Childbirth within the last 6 months
16. Neurological disorders known to affect continence, including spinal cord injury, advanced multiple sclerosis or Parkinson's disease and debilitating stroke
17. Chronic abdominal pain in the absence of diarrhea
18. Presence of an active (turned on) sacral neuromodulator within the last 6 months
19. Pelvic floor surgery (including anal sphincteroplasty) within the past 6 months.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject must have a vagina
Enrollment: 31 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
St. Mark's Incontinence Score | Baseline to 10 weeks
  Validated survey of fecal incontinence severity, score ranges from 0-24, Higher scores indicate more severe symptoms

SECONDARY OUTCOMES:
Change in Fecal incontinence episodes | Baseline to 10 weeks
  Percent improvement= number of fecal incontinence episodes at 10 weeks divided by the number of incontinence epsiodes at baseline.
Fecal Incontinence Quality of Life Scale (FIQoL) | Change in score from baseline to 10 weeks
  Validated Survey evaluates four areas- coping, depression, lifestyle and embarrassment. Each area is scored from 1-5. Higher numbers indicate more severe symptoms. Area scores are not combined
Cumulative adherence correlation with change in St. Mark's score | baseline to 10 weeks
  Adherence as a percentage of all expected exercise sessions (140) correlation with change in St Mark's Incontinence Score (1-24)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Richter, MD PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No